CLINICAL TRIAL: NCT03167593
Title: Evaluation of the Effects of Consumption of the Probiotic Strain Lactobacillus Coryniformis CECT5711 on the Immune Response to Influenza Vaccine in Adults Over 65 Years of Age.
Brief Title: Effects of Lactobacillus Coryniformis CECT5711 on Immune Response to Influenza Vaccination in Adults Over 65.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P039
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Influenza Vaccination; Immune Response; Probiotics
Keywords: Lactobacillus coryniformis; Flu; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Control (Placebo Comparator): Capsules containing 300 mg of maltodextrin.
  Interventions: Other: Control placebo
- Probiotic (Experimental): Capsules containing 3x10(9) colon-forming units of the strain L. coryniformis K8 CECT5711 in a matrix of maltodextrin.
  Interventions: Dietary Supplement: Lactobacillus coryniformis K8 CECT5711

INTERVENTIONS:
Dietary Supplement: Lactobacillus coryniformis K8 CECT5711 — Lactobacillus coryniformis CECT5711
  Other Names: Probiotic group
  Arms: Probiotic
Other: Control placebo — Maltodextrin
  Arms: Control

SUMMARY:
The objective of the present study is to evaluate the capability of the probiotic strain Lactobacillus coryniformis K8 CECT5711 (Lc K8) to enhance the immune response to influenza vaccine in elderly and the effect on respiratory symptoms related to respiratory infections.

A randomized, double-blind, placebo-controlled trial was conducted between November of 2015 and April of 2016. A total of 98 residents of nursing homes aged more than 65 years were randomly assigned to receive Lc K8 or placebo for two weeks previous to influenza vaccination.

Primary outcome was the percentage of seroconversion. Secondary outcome were the incidence of influenza-like illness and respiratory symptoms associated to respiratory infections during the follow-up period of 5 months. Serum cytokines and immunoglobulins levels were also evaluated.

DETAILED DESCRIPTION:
The objective of the present study is to evaluate the capability of Lc K8 to enhance the immune response to influenza vaccine in elderly and the effect on respiratory symptoms related to respiratory infections.

A randomized, double-blinded, placebo controlled, multicenter trial was performed. The study was started on October 2015 and ended on April 2016. The recruitment of volunteers was carried out in five nursing home of Granada (Spain) at the beginning of the vaccination program.

Volunteers were randomly assigned to one of two groups. Those in the placebo group daily consumed a capsule containing 300 mg of maltodextrin. Those in the probiotic group daily consumed a capsule containing 3x10(9) colon-forming units of the strain Lc K8 in a matrix of maltodextrin.

From two weeks previous to the beginning of the intervention the consumption of any probiotic supplement was restricted until the end of the study. During two weeks before flu vaccination volunteers daily received a capsule of probiotic or placebo. Day 15 of the study all volunteers received intramuscular vaccination against flu (inactivated trivalent influenza: A/California/7/22009[H1N1]pdm09, A/HongKong/4801/2014[H3N2], B/Brisbane/60/2002) for the vaccine campaign of 2015/2016 (Sanofi Pasteur Europe, Lyon, France). All volunteers were vaccinated during the same week (second week of November 2015). After vaccination volunteer were followed-up until 31 of April 2016.

ELIGIBILITY:
Inclusion Criteria:

* Residents in nursing home aged more than 65 years

Exclusion Criteria:

* Frequent gastrointestinal diseases, antibiotic treatment during the intervention, allergy to any groups of antibiotics, egg proteins or adjuvants and excipients of the flu vaccine

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-10-01; Primary Completion 2016-01-07 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of seroconversion | 2 months
  According to the European Centre for Disease Prevention and Control (ECDC) for population older than 60 years old, seroconversion corresponds to the proportion of vaccinated individuals achieving a haemagglutination-inhibition (HAI) titre of >1:40 or a significant increase in HAI antibody titre, i.e. at least a four-fold titre increase.

SECONDARY OUTCOMES:
Incidence of influenza-like illness | 5 months
  Number of cases of influenza-like illness during the follow-up period (5 months)

OTHER OUTCOMES:
Cytokines | 3 months
  Interleukin-10, interleukin-4, tumor necrosis factor -alpha
Immunoglobulins | 3 months
  Immunoglobulin A (IgA) and Immunoglobulin G (IgG)
Gastrointestinal manifestations | 5 months
  Nausea, vomits and lack of appetite during follow-up period
Medication | 5 months
  Consumption of analgesics and antibiotics during follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gracián, MD, Principal Investigator — Hospital de San Rafael, Granada (Spain)

IPD SHARING:
Plan to Share IPD: No